CLINICAL TRIAL: NCT05472506
Title: A Phase 1b, Open-Label, Single-Arm Dose-Expansion Study of IK-175, an Oral Aryl Hydrocarbon Receptor Inhibitor, in Combination With Nivolumab in Patients With Primary PD-1 Inhibitor Resistant Metastatic or Locally Incurable, Recurrent HNSCC
Brief Title: Oral AHR Antagonist in Combination With Nivolumab in Patients With PD-1 Resistant Metastatic or Recurrent Head and Neck Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Ikena Oncology (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IK175-002
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer; Head Cancer; Neck Cancer; Head Cancer Neck; Neck Carcinoma
Keywords: IK-175; AHR antagonist; AHR inhibitor; Aryl Hydrocarbon Receptor Antagonist; Immunooncology; AHRi; Aryl Hydrocarbon Receptor Inhibitor; Antagonist; Inhibitor; anti-PD1; aPD1; nivolumab; checkpoint inhibitor; CPI; combination therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to Cohort 1 or Cohort 2
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): 600 mg qd PO IK-175 + nivolumab
  Interventions: Drug: IK-175 + nivolumab
- Cohort 2 (Experimental): 450 mg q12h PO IK-175 + nivolumab
  Interventions: Drug: IK-175 + nivolumab

INTERVENTIONS:
Drug: IK-175 + nivolumab — IK-175 + nivolumab

SUMMARY:
This is a phase 1b study in adult patients diagnosed with resistant or recurrent head and neck squamous cell carcinoma (HNSCC) designed to assess the safety and tolerability of IK-175 in combination with nivolumab. Disease response, pharmacokinetics (PK), pharmacodynamics, and response biomarkers will also be assessed.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase 1b dose-expansion study to evaluate the safety, tolerability, preliminary antitumor activity, PK, and pharmacodynamics of 2 dose levels of IK-175, administered PO in combination with nivolumab, in patients with primary PD-1-resistant metastatic or locally incurable, recurrent HNSCC for which standard therapy is no longer effective or is intolerable.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Subject has a histologically confirmed metastatic or locally incurable, recurrent HNSCC that has progressed within 12 weeks of initiation of PD-1 inhibitor agent, whether it was administered alone or in combination with chemotherapy.
* Tumors must express PD-L1 with a minimum CPS ≥ 1.
* Subjects can be enrolled regardless of their tumor's expression of human papillomavirus (HPV).
* Subjects are required to have received prior treatment with a platinum-based chemotherapy in the recurrent or metastatic disease setting, unless medically contraindicated.
* Subject has at least 1 measurable lesion per RECIST v1.1.

Key Exclusion Criteria:

* Subject has untreated or symptomatic central nervous system (CNS) tumors or brain metastases.
* Subject must have recovered to ≤ Grade 1 from clinically significant AEs related to prior therapy (eg, myelosuppression or renal or hepatic dysfunction.)
* Subject has received prior treatment with an AHR inhibitor.
* Subject has a medical condition that limits oral administration or impairment of gastrointestinal function that is expected to significantly reduce the absorption of IK-175.
* Uncontrolled or life-threatening symptomatic concomitant disease.
* Clinically significant cardiovascular disease as defined in the protocol.
* Subject is on a medication that is a sensitive substrate of CYP2C8, 2C9, 2C19, or 3A4 that cannot be substituted.
* Females who are pregnant or breastfeeding.

Other inclusion/exclusion criteria are listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs) in subjects receiving IK-175 in combination with nivolumab [Safety and Tolerability] | Treatment Period (Approximately 18 months)
  Number and severity of TEAEs as assessed by CTCAE 5.0
Frequency and severity of treatment related adverse events (TRAEs) in subjects receiving IK-175 in combination with nivolumab [Safety and Tolerability] | Treatment Period (Approximately 18 months)
  Number and severity of TRAEs as assessed by CTCAE 5.0
Frequency and severity of serious adverse events (SAEs) in subjects receiving IK-175 in combination with nivolumab [Safety and Tolerability] | Treatment Period (Approximately 18 months)
  Number and severity of SAEs as assessed by CTCAE 5.0
Frequency and severity of adverse events leading to dose modifications and/or treatment discontinuation in subjects receiving IK-175 in combination with nivolumab [Safety and Tolerability] | Study Treatment Period (Approximately 18 months)
  Number and severity of adverse events leading to dose modifications and/or treatment discontinuation as assessed by CTCAE 5.0
Preliminary antitumor activity of IK-175 treatment in combination with nivolumab: Objective response rate (ORR) | Through study completion including the Treatment Period (approximately 18 months) and the Follow-Up Period (Up to 6 months)
  ORR is defined as the percentage of participants with confirmed complete response (cCR) or confirmed partial response (cPR) per RECIST 1.1
Preliminary antitumor activity of IK-175 treatment in combination with nivolumab: Disease control rate (DCR) | Through study completion including the Treatment Period (approximately 18 months) and the Follow-Up Period (Up to 6 months)
  DCR is defined as the percentage of participants with no occurrence of progressive disease with either cCR, cPR, or stable disease [SD] ≥ 16 weeks per RECIST 1.1 from the beginning of study therapy
Preliminary antitumor activity of IK-175 treatment in combination with nivolumab: Duration of response (DOR) | Through study completion including the Treatment Period (approximately 18 months) and the Follow-Up Period (Up to 6 months))
  DOR is defined as the time from the first documented CR or PR per RECIST 1.1 until disease progression or death from any cause

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of IK-175 when administered in combination with nivolumab: half-life (t1/2) | Time Frame: Day 1, 2, 15 of Cycle 1, Day 1 of Cycles 2-3 (every 28 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 56 days) through end of treatment (approximately 18 months)
  Determine IK-175 half-life (t1/2)
PK of IK-175 when administered in combination with nivolumab: area under the plasma concentration-time curve (AUC) | Time Frame: Day 1, 2, 15 of Cycle 1, Day 1 of Cycles 2-3 (every 28 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 56 days) through end of treatment (approximately 18 months)
  Determine IK-175 AUC
PK of IK-175 when administered in combination with nivolumab: maximum serum concentration (Cmax) | Time Frame: Day 1, 2, 15 of Cycle 1, Day 1 of Cycles 2-3 (every 28 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 56 days) through end of treatment (approximately 18 months)
  Determine IK-175 Cmax
PK of IK-175 when administered in combination with nivolumab: minimum serum concentration (Cmin) | Time Frame: Day 1, 2, 15 of Cycle 1, Day 1 of Cycles 2-3 (every 28 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 56 days) through end of treatment (approximately 18 months)
  Determine IK-175 Cmin
Preliminary antitumor activity of IK-175 in combination with nivolumab: Progression-free survival (PFS) median and at 6 months | Through study completion including the Treatment Period (approximately 18 months) and the Follow-Up Period (Up to 6 months)
  PFS is defined as the length of time from the beginning of study treatment to the first observed disease progression or death due to any cause
Preliminary antitumor activity of IK-175 in combination with nivolumab: Overall survival (OS), median and at 6 months | Through study completion including the Treatment Period (approximately 18 months) and the Follow-Up Period (Up to 12 months)
  OS is defined as the length of time from the beginning of study treatment to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Kim, MD, Study Director — Ikena Oncology; Karim Malek, MD, Study Chair — Ikena Oncology
Locations (4):
- United States (4):
  - University of Chicago Medical Center, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No